CLINICAL TRIAL: NCT05890105
Title: A Phase 1, Randomized, Double-Blind, Sponsor-Open, Placebo-Controlled, Crossover, First-in-Human Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Oral Doses of PF-07853578 Administered to Healthy Adult Participants
Brief Title: A Study to Learn About the Study Medicine PF-07853578 and How it Acts in the Bodies of Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: C5161001
Record Dates: First submitted 2023-05-25; First posted 2023-06-06 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Single dose administration of PF-07853578 and placebo. Participants will receive up to 4 dose levels of PF-07853578 and up to 2 dose levels of matching placebo.
  Interventions: Drug: PF-07853578; Drug: Placebo
- Cohort 2 (Experimental): Single dose administration of PF-07853578 and placebo. Participants will receive up to 4 dose levels of PF-07853578 and up to 2 dose levels of matching placebo.
  Interventions: Drug: PF-07853578; Drug: Placebo
- Cohort 3 (Experimental): Single dose administration of PF-07853578 and placebo. Participants will receive up to 4 dose levels of PF-07853578 and up to 2 dose levels of matching placebo.
  Interventions: Drug: PF-07853578; Drug: Placebo

INTERVENTIONS:
Drug: PF-07853578 — PF-07853578 will be administered as oral solutions or suspensions as escalating single doses to be determined.
Drug: Placebo — Placebo will be administered as oral solutions or suspensions as escalating single doses to be determined.

SUMMARY:
The purposes of this study are:

* To see how the new medicine (PF-07853578) under study is tolerated. And if there are any important side effects. And, how people feel after taking single increasing amount of the medicine by mouth.
* To measure the amount of study medicine in your blood after the medicine is taken by mouth.

This study is seeking for participants who:

* are females of 18 to 65 years old and are not able to give birth to a child.
* are males of 18 to 65 years old.
* have body mass index of 16 to 31 kilograms per meter squared.
* have a total body weight of more than 50 kilograms (110 pounds). Participants will be randomly selected to receive either study medicine (PF-07853578) or placebo (a pill that has no medicine in it). Participants may receive up to 4 amounts of study medicine and up to 2 amounts of placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants of non-childbearing potential and male participants aged 18 to 65 years at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
2. BMI of 16 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention, with the exception of moderate or strong cytochrome P450 3A (CYP3A) inducers or inhibitors which are prohibited within 14 days plus 5 half-lives prior to the first dose of study intervention.
3. Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer). Participation in studies of other investigational products (drug or vaccine) at any time during their participation in this study.
4. Screening supine blood pressure (BP) ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic) for participants <60 years; and ≥150/90 mm/Hg for participants ≥60 years old, following at least 5 minutes of supine rest.
5. Renal impairment as defined by an estimated glomerular filtration rate (eGFR) of <75 mL/min/1.73m².
6. Hematuria as defined by >1+ heme on urine dipstick.
7. Albuminuria as defined by albumin/creatine (Cr) ratio on spot urine albumin (UA) >30 mg/g.
8. Standard 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.
9. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

   * Alanine aminotransferase (ALT), aspartate aminotransferase (AST), Bilirubin ≥1.05×ULN.
   * Total cholesterol, triglycerides, or direct LDL ≥1.25×ULN.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - New Haven Clinical Research Unit, New Haven, Connecticut
  - Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5161001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 23 participants were enrolled, and received at least 1 dose of study intervention.
Groups:
- Cohort 1: Cohort 1 included 4 sequences, each sequence of which included 4 treatment periods: Placebo Fasted->PF-07853578 10 mg [10 mg]->100 mg->500 mg; 1 mg (low dosage strength [LDS])->Placebo Fasted->100 mg->500 mg; 1 mg (LDS)->10 mg->Placebo Fasted->500 mg; and 1 mg (LDS)->10 mg->100 mg->Placebo Fasted
- Cohort 2: Cohort 2 included 4 sequences, each sequence of which included 4 treatment periods: Placebo Fasted->30 mg->300 mg->300 mg Fed; 3 mg->Placebo Fasted->300 mg->300 mg fed; 3 mg->30 mg->Placebo Fasted->Placebo Fed; and 3 mg->30 mg->300 mg->300 mg fed
- Cohort 3: Cohort 3 included 2 sequences, each sequence of which included 2 treatment periods: Placebo Fasted->Placebo Fasted; and 8 mg->8 mg (intermediate dosage strength [IDS])
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 8 | 8 | 7
Completed | 6 | 6 | 7
Not Completed | 2 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Other | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 8 | 8 | 7 | 23
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 6 | 5 | 6 | 17
  45-64 years | 2 | 3 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2
  Male | 7 | 7 | 7 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 7 | 7 | 6 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 4 | 1 | 8
  Black or African American | 3 | 2 | 5 | 10
  Asian | 2 | 1 | 1 | 4
  American Indian or Alaska Native | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An adverse event is considered a TEAE if the event started during the effective duration of treatment. All events that started on or after the first dosing day and time/start time, if collected, but before the end of the study were flagged as TEAEs. The algorithm did not consider any events that started prior to the first dose date. Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Day 1-11 in each period, along with the 29-36 day post final dose follow-up
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received.
Measure: Count of Participants; unit: Participants
Groups:
- PF-07853578 1 mg (1mg) (Low Dosage Strength [LDS] Solution): Participants in Cohort 1 received 1 mg (LDS Solution).
- 3 mg: Participants in Cohort 2 received 3 mg.
- 8 mg: Participants in Cohort 3 received 8 mg.
- 8 mg (Intermediate Dosage Strength [IDS] Solution): Participants in Cohort 3 received 8 mg (IDS Solution)
- 10 mg: Participants in Cohort 1 received 10 mg.
- 30 mg: Participants in Cohort 2 received 30 mg.
- 100 mg: Participant in Cohort 1 received 100 mg.
- 300 mg: Participants in Cohort 2 received 300 mg.
- 300 mg Fed: Participants in Cohort 2 received 300 mg Fed.
- 500 mg: Participants in Cohort 1 received 500 mg.
- Placebo Fasted: Participants in Cohorts 1, 2, and 3 received Placebo Fasted.
- Placebo Fed: Participants in Cohort 2 received Placebo Fed.
Arm/Group | PF-07853578 1 mg (1mg) (Low Dosage Strength [LDS] Solution) | 3 mg | 8 mg | 8 mg (Intermediate Dosage Strength [IDS] Solution) | 10 mg | 30 mg | 100 mg | 300 mg | 300 mg Fed | 500 mg | Placebo Fasted | Placebo Fed
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 5 | 6 | 5 | 6 | 5 | 4 | 14 | 1
Participants
  All-causality AEs | 1 | 2 | 3 | 2 | 2 | 1 | 0 | 1 | 4 | 0 | 3 | 0
  Treatment-related AEs | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  All-causality SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Treatment-related SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities Meeting Pre-Defined Categorical Criteria Without Regard to Baseline Abnormality
Description: Pre-defined categorical criteria for laboratory abnormalities included: Lymphocytes <0.8 x lower limit of normal (LLN); Basophils/Leukocytes > 1.2 x upper limit of normal (ULN); Eosinophils/Leukocytes >1.2 x ULN; Monocytes/Leukocytes >1.2 x ULN; low-density lipoprotein (LDL) Direct Endpoint Measure >1.2 x ULN; Triglycerides >1.3 x ULN; Specific Gravity <1.003 or >1.030; pH >8; Ketones ≥1; Urobilinogen (EU) ≥1; URINE Bilirubin ≥1; Leukocyte Esterase ≥1.
Time Frame: Day 1-11 in each period, along with the 29-36 day post final dose follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07853578 1 mg (1mg) (Low Dosage Strength [LDS] Solution) | 3 mg | 8 mg | 8 mg (Intermediate Dosage Strength [IDS] Solution) | 10 mg | 30 mg | 100 mg | 300 mg | 300 mg Fed | 500 mg | Placebo Fasted | Placebo Fed
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 5 | 6 | 5 | 6 | 5 | 4 | 14 | 1
Participants | 4 | 5 | 5 | 4 | 5 | 5 | 4 | 4 | 2 | 1 | 11 | 1

3. Primary Outcome: Number of Participants With Vital Signs Abnormalities Meeting Pre-Defined Categorical Criteria
Description: Vital signs categorical criteria: 1) supine systolic blood pressure (SBP) <90 millimeters of mercury (mmHg); 2) supine diastolic blood pressure (DBP) <50 mmHg; 3) supine pulse rate <40 or >120 beats per minute (bpm); 4) change from baseline (increase or decrease) in supine SBP greater than or equal to (≥) 30 mmHg; 5) change from baseline (increase or decrease) in supine DBP ≥ 20 mmHg.
Time Frame: Day 1-11 in each period, along with the 29-36 day post final dose follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07853578 1 mg (1mg) (Low Dosage Strength [LDS] Solution) | 3 mg | 8 mg | 8 mg (Intermediate Dosage Strength [IDS] Solution) | 10 mg | 30 mg | 100 mg | 300 mg | 300 mg Fed | 500 mg | Placebo Fasted | Placebo Fed
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 5 | 6 | 5 | 6 | 5 | 4 | 14 | 1
Participants
  DBP <50 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Pulse rate < 40 bpm | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate > 120 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP <90 mmHg | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
  Change from baseline in DBP ≥20 increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Change from baseline in DBP ≥20 decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Change from baseline in SBP ≥30 mmHg increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Change from baseline in SBP ≥30 mmHg decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

4. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Meeting Pre-Defined Categorical Criteria
Description: ECG categorical criteria: 1. PR interval (the interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization): a) ≥300 millisecond (msec), b) ≥25% increase when baseline is > 200 msec, c) ≥50% increase when baseline is less than or equal to (≤) 200 msec.
  2. QRS interval (time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization): a) ≥140 msec, b) ≥50% increase from baseline.
  3. QTcF interval (QT corrected using the Fridericia formula): a) >450 msec and ≤480 msec, b) >480 msec and ≤500 msec, c) >500 msec, d) >30 msec and ≤60 msec increase from baseline, e) >60 msec increase from baseline.
Time Frame: Day 1-11 in each period, along with the 29-36 day post final dose follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07853578 1 mg (1mg) (Low Dosage Strength [LDS] Solution) | 3 mg | 8 mg | 8 mg (Intermediate Dosage Strength [IDS] Solution) | 10 mg | 30 mg | 100 mg | 300 mg | 300 mg Fed | 500 mg | Placebo Fasted | Placebo Fed
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 5 | 6 | 5 | 6 | 5 | 4 | 14 | 1
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Maximum Concentration Observed in Plasma (Cmax)
Description: Maximum observed plasma PF-07328948 concentration. Observed directly from data.
Time Frame: Pre-dose (0 hour) and 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours and 12 hours post Day 1 dosing of each treatment period (Periods 1-4)
Population: All participants randomly assigned to study intervention and who received at least 1 dose of study intervention and had at least 1 of the PK parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-07853578 1 mg (1mg) (Low Dosage Strength [LDS] Solution) | 3 mg | 8 mg | 8 mg (Intermediate Dosage Strength [IDS] Solution) | 10 mg | 30 mg | 100 mg | 300 mg | 300 mg Fed | 500 mg
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 5 | 6 | 5 | 6 | 5 | 4
nanogram per milliliter (ng/mL) | 7.196 (14) | 7.226 (52) | 14.87 (66) | 41.92 (41) | 17.92 (35) | 43.91 (45) | 119.8 (38) | 355.6 (39) | 690.6 (53) | 449.2 (51)

6. Secondary Outcome: Time to Achieve Cmax (Tmax)
Description: Observed directly from data as time of first occurrence.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | PF-07853578 1 mg (1mg) (Low Dosage Strength [LDS] Solution) | 3 mg | 8 mg | 8 mg (Intermediate Dosage Strength [IDS] Solution) | 10 mg | 30 mg | 100 mg | 300 mg | 300 mg Fed | 500 mg
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 5 | 6 | 5 | 6 | 5 | 4
hours (hr) | 0.500 [0.500 to 1.00] | 1.08 [0.500 to 1.17] | 1.00 [0.500 to 1.00] | 0.517 [0.500 to 0.517] | 1.00 [0.500 to 2.00] | 2.00 [1.00 to 2.00] | 3.00 [2.00 to 3.02] | 2.00 [1.00 to 3.00] | 4.00 [2.00 to 6.00] | 3.02 [2.00 to 6.00]

7. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Measured Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration. It was determined by using linear/Log trapezoidal method.
Time Frame: Pre-dose (0 hours) and 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours and 12 hours post Day 1 dosing of each treatment period (Periods 1-4)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-07853578 1 mg (1mg) (Low Dosage Strength [LDS] Solution) | 3 mg | 8 mg | 8 mg (Intermediate Dosage Strength [IDS] Solution) | 10 mg | 30 mg | 100 mg | 300 mg | 300 mg Fed | 500 mg
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 5 | 6 | 5 | 6 | 5 | 4
nanogram*hour per milliliter (ng*hr/mL) | 17.03 (30) | 43.52 (77) | 105.8 (62) | 111.6 (44) | 153.3 (33) | 462.4 (54) | 1825 (31) | 4590 (58) | 6747 (66) | 7774 (25)

8. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Extrapolated Infinite Time (AUCinf)
Description: Area under the plasma concentration-time curve from time 0 extrapolated to infinite time. AUCinf = AUClast + (Clast*/kel), where Clast* was the predicted plasma concentration at the last quantifiable timepoint estimated from the log-linear regression analysis, and Kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve, AUClast = Area under the plasma concentration time-curve from zero to the last measured concentration.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-07853578 1 mg (1mg) (Low Dosage Strength [LDS] Solution) | 3 mg | 8 mg | 8 mg (Intermediate Dosage Strength [IDS] Solution) | 10 mg | 30 mg | 100 mg | 300 mg | 300 mg Fed | 500 mg
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 5 | 6 | 5 | 6 | 5 | 4
ng*hr/mL | 18.29 (31) | 46.69 (73) | 111.5 (60) | 114.1 (44) | 157.0 (33) | 470.6 (55) | 1876 (29) | 4649 (59) | 6822 (67) | 8066 (27)

9. Secondary Outcome: Terminal Half-Life (t1/2)
Description: Terminal elimination half-life. t1/2 = Loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Only those data points judged to describe the terminal log linear decline were used in the regression.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours (hr)
Arm/Group | PF-07853578 1 mg (1mg) (Low Dosage Strength [LDS] Solution) | 3 mg | 8 mg | 8 mg (Intermediate Dosage Strength [IDS] Solution) | 10 mg | 30 mg | 100 mg | 300 mg | 300 mg Fed | 500 mg
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 5 | 6 | 5 | 6 | 5 | 4
hours (hr) | 5.748 (4.1227) | 12.78 (3.6983) | 15.19 (7.1273) | 8.692 (2.4278) | 11.26 (4.7825) | 13.15 (2.5990) | 13.00 (3.8601) | 10.44 (2.7311) | 11.28 (2.7070) | 14.38 (3.0237)

ADVERSE EVENTS:
Time Frame: Day 1-11 in each period, along with the 29-36 day post final dose follow-up
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | PF-07853578 1 mg (1mg) (Low Dosage Strength [LDS] Solution) | 3 mg | 8 mg | 8 mg (Intermediate Dosage Strength [IDS] Solution) | 10 mg | 30 mg | 100 mg | 300 mg | 300 mg Fed | 500 mg | Placebo Fasted | Placebo Fed
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/5 | 0/5 | 0/5 | 0/6 | 0/5 | 0/6 | 0/5 | 0/4 | 0/14 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/5 | 0/5 | 0/5 | 0/6 | 0/5 | 0/6 | 0/5 | 0/4 | 0/14 | 0/1
Other Adverse Events (participants affected / at risk) | 1/5 | 2/6 | 3/5 | 2/5 | 2/5 | 1/6 | 0/5 | 1/6 | 4/5 | 0/4 | 3/14 | 0/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-07853578 1 mg (1mg) (Low Dosage Strength [LDS] Solution) (N=5) | 3 mg (N=6) | 8 mg (N=5) | 8 mg (Intermediate Dosage Strength [IDS] Solution) (N=5) | 10 mg (N=5) | 30 mg (N=6) | 100 mg (N=5) | 300 mg (N=6) | 300 mg Fed (N=5) | 500 mg (N=4) | Placebo Fasted (N=14) | Placebo Fed (N=1)
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Application site irritation (General disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Feeling hot (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Any untoward findings identified on physical and/or neurological examinations, and cardiac monitoring conducted during the active collection period were captured as adverse events, if those findings met the definition of an AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/05/NCT05890105/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT05890105/SAP_001.pdf